CLINICAL TRIAL: NCT04064424
Title: Cancer Prevention & Online Technologies
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB-50303; IRB-50303 (Other: Stanford-IRB); SKIN0049 (Other: OnCore); 1DP2CA225433-01 (NIH)
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Skin Cancer
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention Advertisement (Experimental): Participants will be exposed to prevention videos and images through Facebook Advertising
  Interventions: Other: Prevention video advertisement; Other: Prevention images for advertisement
- No Advertisement (Active Comparator): No prevention videos and images will be shown through Facebook Advertising
  Interventions: Other: No Advertisement

INTERVENTIONS:
Other: Prevention video advertisement — Skin Cancer Prevention videos
  Arms: Prevention Advertisement
Other: Prevention images for advertisement — Skin Cancer Prevention images
  Arms: Prevention Advertisement
Other: No Advertisement — No skin cancer prevention videos or images were advertised.
  Arms: No Advertisement

SUMMARY:
The overall goal of this research is to develop interventions that leverage online technology (e.g. ads, social media) to reduce individuals' skin-cancer-related risk behaviors and ultimately to reduce skin cancer incidence.

DETAILED DESCRIPTION:
This research includes three phases:

1. To better understand the motivators and inhibitors of skin cancer risk behaviors in various populations including use of indoor tanning and outdoor sun exposure;
2. To develop content messages and images related to skin cancer risk that are resonant with various populations;
3. To test the relative effectiveness of these messages in reducing likelihood of or actual skin cancer risk behaviors in various populations.

ELIGIBILITY:
Inclusion Criteria:

* Facebook user between the age of 18 and 65
* Self-identifies as male
* Profile indicates interest in at least one of the following: LGBT community, LGBT culture, LGBT social movements, Rainbow flag, Gay pride, GAY-friendly, homosexuality

Exclusion Criteria:

* Failure to meet inclusion criteria

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 720000 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Measure intent to tan | 4 weeks
  Intent to tan will be measured by our follow-up survey question. Rates of each response will be compared between experimental groups.

SECONDARY OUTCOMES:
Measure awareness of indoor tanning risk | 4 weeks
  Awareness of indoor tanning risk will be measured by our follow-up survey question. Rates of each response will be compared between experimental groups.

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Linos, Principal Investigator — Stanford University

IPD SHARING:
Plan to Share IPD: No